CLINICAL TRIAL: NCT07171710
Title: Comparative Evaluation of 0.05% Cyclosporine A Plus Absorbable Punctal Plugs Versus 0.05% Cyclosporine A Monotherapy in Sjögren's Syndrome-Associated Dry Eye: A Paired-Eye Study
Brief Title: Efficacy of 0.05% Cyclosporine A Eye Drops Combined With Absorbable Tear Duct Plugs in the Treatment of Dry Eye in Sjögren's Syndrom
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zhangyi2024-1
Record Dates: First submitted 2025-09-08; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-10

CONDITIONS: Dry Eye Disease
Keywords: dry eye disease; Absorbable Tear Duct Plugs; Cyclosporine
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Other): One eye was randomized to recieve a Smart plug absorbable lacrimal duct plugs, and cyclosporin A 0.05% cyclosporine A eye drops were administered three times daily to both eyes.
  Interventions: Drug: 0.05% Cyclosporine Eye Drops
- Control group (Other): cyclosporin A 0.05% cyclosporine A eye drops were administered three times daily to both eyes.
  Interventions: Drug: 0.05% Cyclosporine Eye Drops; Device: Smart plug absorbable lacrimal duct plugs

INTERVENTIONS:
Drug: 0.05% Cyclosporine Eye Drops — Cyclosporin A 0.05% eye drops were administered twice daily to both eyes
Device: Smart plug absorbable lacrimal duct plugs — The lacrimal duct embolization implant is performed by partially sealing the tear discharge duct to increase the lubrication of natural tears on the eye surface.
  Arms: Control group

SUMMARY:
To study the effectiveness of 0.05% cyclosporine A eye drops in combination with smart plug absorbable lacrimal duct plugs in the monotherapy of cyclosporine for SSDE.

DETAILED DESCRIPTION:
Participants meeting all eligibility criteria were enrolled and randomized to receive combined treatment (0.05% cyclosporine A plus absorbable punctal plug) in one eye and 0.05% cyclosporine A monotherapy in the contralateral eye. Eye allocation (left or right) was determined using block randomization with a fixed block size of two, implemented via an online randomization tool (www.sealedenvelope.com). The randomization sequence was generated in advance by an independent biostatistician who was not involved in patient care or data analysis.

Treatment allocation was concealed using sequentially numbered, opaque, sealed envelopes (SNOSE), which were prepared by an independent biostatistician not involved in patient care or outcome assessment. At the time of enrollment, a study coordinator opened the next envelope in sequence to determine which eye would receive the combined treatment. The contralateral eye automatically received cyclosporine A monotherapy.

To maintain masking, the ophthalmologists responsible for outcome assessment (including ocular surface staining, tear film measurements, and in vivo confocal microscopy) were blinded to the treatment allocation. Participants were informed that both eyes would receive active treatment and were not informed of the specific allocation. The investigators performing plug insertion and administering cyclosporine A were not involved in any clinical evaluations.

A total of 30 patients with Sjögren's syndrome-associated dry eye (SSDE) were planned for enrollment. The sample size calculation was based on a paired-eye design, in which each participant served as their own control. The calculation assumed a two-sided significance level of 0.05 (α = 0.05) and a statistical power of 95% (β = 0.05), aiming to detect a clinically meaningful difference in ocular surface parameters (e.g., tear breakup time or symptom scores) between the two eyes. The estimated required sample size accounted for potential dropouts and was deemed sufficient to identify within-subject differences while minimizing variability due to inter-individual factors such as disease severity, lifestyle, and systemic autoimmune status.

ELIGIBILITY:
Inclusion Criteria:

1. The patients aged ≥18 years who had a confirmed diagnosis of Sjögren's syndrome (SS).
2. Dry eye diagnosis required both subjective and objective criteria: participants presented with one or more ocular surface symptoms such as dryness, foreign body sensation, burning, fatigue, discomfort, redness, or fluctuating vision, with an Ocular Surface Disease Index (OSDI) score of ≥13; Noninvasive Tear Break-Up Time (NIBUT)≤10s and Schirmer I test≤ 5 mm/5 min
3. voluntarily participate in this study and sign written informed consent

Exclusion Criteria:

1. Any patient with structural abnormalities (eyelid scars, entropion, trichiasis, etc.);
2. Patients with any inflammation or active structural changes in the iris or anterior chamber;
3. Glaucoma;
4. Patients who have undergone previous ophthalmic surgery or have undergone timely closure;
5. Patients using any topical medications other than artificial tears, 0.1% flumirone eye drops, and 0.05% cyclosporine A eye drops;
6. Patients who received any systemic or topical antibacterial or anti-inflammatory drug treatment 90 days before the start of the study;
7. Patients wearing contact lenses;
8. Patients with corneal infection;
9. Corneal diseases (marginal ulcers, opacity, scars, bullous keratopathy, conjunctival laxity, eyelid ball adhesions or tumors);
10. Pregnancy;
11. Study the changes of immunosuppressive system treatment in the first 90 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The Ocular Surface Disease Index (OSDI) score | Assessed after 3 months of the trial
  The Ocular Surface Disease Index (OSDI) is a tool used for screening and diagnosing patients with dry eye syndrome. It assesses the severity of dry eye, covering three dimensions: ocular symptoms, visual function and environmental triggers
VAS score | Assessed after 3 months of the trial
  A swimming ruler of about 10cm in length was used, with 10 scales on one side and "0" and "10" ends, respectively, with 0 indicating no pain and 10 indicating the most severe pain that was unbearable.
BUT | Assessed after 6 months of the trial
  Tear film break-up time,It is a tear stability test
tear river height | Assessed after 6 months of the trial
  The concave arc formed at the junction of tears and eyelid margin was observed under a slit lamp microscope, and the tear secretion was indirectly evaluated by measuring the tear retention height
IVCM examination | Assessed after 6 months of the trial
  It can observe the physiological and pathological changes of ocular surface tissues and cell structures in vivo, and has wide applications in the diagnosis and treatment evaluation of infectious keratitis, ocular surface assessment of dry eye disease, evaluation of the therapeutic effect of ocular surface surgery, and early screening of diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Study Director — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Dong Y, Cao JF, Li ZC, Yang XY, Chen L. Enhanced efficacy of 0.05% cyclosporine a combined with absorbable punctal plugs in Sjogren's syndrome-associated dry eye: a paired-eye clinical trial. Front Med (Lausanne). 2026 Jan 6;12:1674647. doi: 10.3389/fmed.2025.1674647. eCollection 2025. PMID 41567664